CLINICAL TRIAL: NCT04506853
Title: Single-Sided Deafness and Asymmetric Hearing Loss Post-Approval Study
Brief Title: Single-Sided Deafness and Asymmetric Hearing Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P000025/S113
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Unilateral; Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Procedure (Other)
  Interventions: Device: MED-EL Cochlear Implant System

INTERVENTIONS:
Device: MED-EL Cochlear Implant System — Cochlear implant and audio processor

SUMMARY:
The purpose of the study is to evaluate the long-term safety and effectiveness of cochlear implantation of the approved population in adults and children with single-sided deafness and asymmetric hearing loss.

DETAILED DESCRIPTION:
The study will be conducted as a single-subject, repeated measures, multi center study at 6 sites. Sixty-five subjects will be enrolled in this study. Six centers across the United States and Canada will recruit subjects into this study. Study subjects will be followed for a minimum of 3 years post-implantation of the device.

ELIGIBILITY:
Inclusion Criteria:

* Five years of age or older at the time of implantation
* Unilateral profound hearing loss, as defined by a pure-tone average (500, 1000, 2000, and 4000 Hz) of 90 dB or greater in the ear to be implanted
* Sensorineural hearing loss in the ear to be implanted, as defined by an air-bone gap less than or equal to 10 dB at two or more frequencies out of 500, 1000, 2000, and 4000 Hz and a diagnosed pathology of the outer or middle ear
* Normal hearing or mild to moderate hearing loss in the non-implanted ear, as defined by a pure-tone average (500, 1000, 2000, and 4000 Hz) of 55 dB or less
* Word recognition in the ear to be implanted of 5% or less on CNC word score in quiet
* Previous experience with an appropriately-fit Contralateral Routing of Signal (CROS) hearing aid, BI-Contralateral Routing of Signal (CROS) hearing aid, bone conduction, or traditional hearing aid, as deemed appropriate by investigator
* Fluent in English

Exclusion Criteria:

* Duration of profound hearing loss of 10 years or more
* Absence of cochlear development or non-functionality of cochlear nerve
* Other retrocochlear hearing loss
* Evidence of severe cochlear malformation (i.e., common cavity or ossification)
* External or middle ear infection
* Suspected developmental or cognitive concern
* Other medical contraindication for surgery or anesthesia

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Long-term performance of the Cochlear Implant System will be assessed through speech perception testing in noise completed through three years (36 months) post implantation | Three years (36 months) post implantation
  The primary effectiveness endpoint will be change on speech in noise when speech is presented to the front and noise is presented to the acoustic hearing (contralateral) ear. The pre-operative, best-aided score will be compared to the 12-month and 36-month CI score for AzBio sentences in noise(range of score 0-100, higher score is better). Improvement is defined as greater than or equal to 10 percentage points.

SECONDARY OUTCOMES:
Long term performance of the Cochlear Implant System will be summarized through speech perception testing in noise completed through three years (36 months) post implantation | Three years (36 months) post implantation
  Speech in noise in two spatial conditions will demonstrate similar performance from the pre-operative, best-aided score to the CI score at 12 and 36 months post-activation. AzBio sentence in noise score will be summarized for two conditions: speech and noise presented from the front as well as speech presented to the front and noise presented to the CI ear.(Range of score 0-100, higher score is better)
Long term performance of the Cochlear Implant System will be assessed through speech perception testing in quiet completed through three (36 months) post implantation | Three years (36 months) post implantation
  Speech perception in quiet will be summarized for the CI ear as well as the contralateral ear at the pre-operative, 12-month, and 36-month intervals. The CI ear is expected to demonstrate improvement (greater than or equal to 10 percentage point change), while the contralateral ear is expected to demonstrate no change. (Range of score 0-100, higher score is better)
Long term subjective benefit of the Cochlear Implant System will be assessed through three years (36 months) post implantation | Three years (36 months) post implantation
  Subjective data will be collected via the Speech, Spatial, and Qualities of Hearing Scale (SSQ). Responses will be summarized from the pre-operative, 12-month, and 36-month intervals.(Range of score 0-10, lower score is better)
Long term safety will be evaluated for all study subjects through three (36 months) years post implantation | Three years (36 months) post implantation
  Safety will be assessed by collecting and reporting device-related adverse events occurring throughout the study. This will be summarized and reported as the number and proportion of subjects experiencing an adverse device event.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - New York Eye and Ear Infirmary, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Virginia Mason Medical Center, Seattle, Washington
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

REFERENCES:
- [Background] Arndt S, Laszig R, Aschendorff A, Hassepass F, Beck R, Wesarg T. Cochlear implant treatment of patients with single-sided deafness or asymmetric hearing loss. HNO. 2017 Aug;65(Suppl 2):98-108. doi: 10.1007/s00106-016-0297-5. PMID 28188428
- [Background] Arndt S, Prosse S, Laszig R, Wesarg T, Aschendorff A, Hassepass F. Cochlear implantation in children with single-sided deafness: does aetiology and duration of deafness matter? Audiol Neurootol. 2015;20 Suppl 1:21-30. doi: 10.1159/000380744. Epub 2015 May 19. PMID 25999052
- [Background] Buss E, Dillon MT, Rooth MA, King ER, Deres EJ, Buchman CA, Pillsbury HC, Brown KD. Effects of Cochlear Implantation on Binaural Hearing in Adults With Unilateral Hearing Loss. Trends Hear. 2018 Jan-Dec;22:2331216518771173. doi: 10.1177/2331216518771173. PMID 29732951
- [Background] Dillon MT, Buss E, Rooth MA, King ER, Deres EJ, Buchman CA, Pillsbury HC, Brown KD. Effect of Cochlear Implantation on Quality of Life in Adults with Unilateral Hearing Loss. Audiol Neurootol. 2017;22(4-5):259-271. doi: 10.1159/000484079. Epub 2018 Jan 4. PMID 29298446
- [Background] Niparko JK, Cox KM, Lustig LR. Comparison of the bone anchored hearing aid implantable hearing device with contralateral routing of offside signal amplification in the rehabilitation of unilateral deafness. Otol Neurotol. 2003 Jan;24(1):73-8. doi: 10.1097/00129492-200301000-00015. PMID 12544032
- [Background] Van de Heyning P, Vermeire K, Diebl M, Nopp P, Anderson I, De Ridder D. Incapacitating unilateral tinnitus in single-sided deafness treated by cochlear implantation. Ann Otol Rhinol Laryngol. 2008 Sep;117(9):645-52. doi: 10.1177/000348940811700903. PMID 18834065
- [Background] Vermeire K, Van de Heyning P. Binaural hearing after cochlear implantation in subjects with unilateral sensorineural deafness and tinnitus. Audiol Neurootol. 2009;14(3):163-71. doi: 10.1159/000171478. Epub 2008 Nov 13. PMID 19005250